CLINICAL TRIAL: NCT01504984
Title: An Open-label, Randomized, Single Dose, Crossover Phase I Clinical Trial to Compare Pharmacokinetic Property of SYO-1126 and Glivec Film Coated Tab., 4T (400mg) in Healthy Male Volunteers
Brief Title: Crossover Study to Compare Pharmacokinetic Property of SYO-1126 and Glivec Film Coated Tab in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Collaborators: Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SYO1126
Record Dates: First submitted 2011-12-27; First posted 2012-01-06 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: Evaluation of the pharmacokinetics equivalence; Healthy volunteers; Single dose over the period I and II(crossover); Healthy male volunteers
MeSH Terms: interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SYO-1126 (Experimental): Imatinib 400mg/tablet, PO, 1 tablet once daily for I&II D1(crossover)
  Interventions: Drug: SYO-1126
- Glivec film coated tab 4T(400mg) (Active Comparator): 100mg/tablet, po, 4 tablets once daily for period I&II D1(crossover)
  Interventions: Drug: Glivec film coated tab 4T(400mg)

INTERVENTIONS:
Drug: SYO-1126 — Imatinib 400mg/tablet, PO, 1 tablet once daily for I&II D1(crossover)
  Other Names: Imatinib 400mg
  Arms: SYO-1126
Drug: Glivec film coated tab 4T(400mg) — Imatinib 100mg/tablet, PO, 4 tablets once daily for period I&II D1(crossover)
  Other Names: Imatinib 100mg; Glivec film coated tab
  Arms: Glivec film coated tab 4T(400mg)

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics equivalence and safety by comparing pharmacokinetics characteristics between the SYO-1126 and Glivec Film Coated tab 4T (400mg) when administered a single-dose to healthy male volunteers.

DETAILED DESCRIPTION:
Healthy volunteers are administrated single-dose over the period I and II (crossover) of SYO-1126 and Glivec Film Coated tab 4T (400mg) as of imatinib 400mg.

Every time before and after each medication, pharmacokinetic (PK) parameters and safety of SYO-1126 and Glivec Film Coated tab 4T (400mg) is performed using a blood sample and conducting some tests (vital signs, physical exam, ECG, laboratory test, etc.) respectively.

ELIGIBILITY:
Inclusion Criteria:

* Between 20aged and 45aged in healthy males
* Over 55kg and BMI: 18.5~25 kg/m2
* Agreement with written informed consent

Exclusion Criteria:

* Subject with symptoms of acute disease at the time of screening
* Clinically significant cardiovascular system, pulmonary system, renal system, endocrine system, blood system, gastrointestinal system, nervous system, mental disease or malignant tumor
* Subject with known for gastrointestinal disease or surgical history which affect on absorption of drug
* An impossible one who participates in clinical trial by result of screening tests
* Inadequate result of laboratory test AST/ALT > 1.5 x UNL Total bilirubin > 1.5 X UNL
* Clinically significant allergic disease(Except for mild allergic rhinitis seems to be not need for medication)
* Subject with known for hypersensitivity reaction to imatinib analog
* Subject with known for history which drug abuse or show positive for it in screening tests
* Previously participate in other trial within 60 days
* Previously make whole blood donation within 60 days or component blood donation within 30 days
* Previously have blood transfusion within 30 days
* Not able to taking the institutional standard meal
* Subject who have had abnormal eating which affect on the ADME of drug
* Not able to taking the grapefruit-containing foods
* Taking ETC(ethical the counter)medicine including oriental medicine within 14 days or taking OTC(over the counter)medicine or vitamin preparations within 7 days
* Continued to be taking caffein(caffein>5cup/day), drinking (alcohol>30g/day) and severe heavy smoker(cigarette>1/2pack/day)
* An impossible one who participates in clinical trial by investigator's decision including for reason laboratory test result

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of the AUCt SYO-1126 anf Glivec Film coated tab 4T(400mg) | 0-72hr
Pharmacokinetics of the Cmax SYO-1126 anf Glivec Film coated tab 4T(400mg) | 0-72hr

SECONDARY OUTCOMES:
Pharmacokinetics of the AUCinf SYO-1126 and Glivec Film Coated 4T(400mg) | 0-72hr
Evaluation of the safety of SYO-1126 and Glivec Film Coated 4T(400mg) from vital signs, physical exam, ECG, laboratory test, adverse events and so on. | 20~24 days
Pharmacokinetics of the Tmax of SYO-1126 and Glivec Film Coated 4T(400mg) | 0-72hr
Pharmacokinetics of the T1/2 of SYO-1126 and Glivec Film Coated 4T(400mg) | 0-72hr
Pharmacokinetics of the CL/F of SYO-1126 and Glivec Film Coated 4T(400mg) | 0-72hr

CONTACTS AND LOCATIONS:
Overall Officials: Min Su Park, Doctor, Principal Investigator — Severance Hospital
Locations (1):
- Severance hospital, Seoul, Seodaemun-gu, South Korea